CLINICAL TRIAL: NCT01823224
Title: A Prospective, Randomized, Double Blind, Comparative-effectiveness Study Comparing Perioperative Administration of Oral Versus Intravenous Acetaminophen for Laparoscopic Cholecystectomy
Brief Title: Comparing Effectiveness of IV vs Oral Acetaminophen Given Perioperatively for Lap Choles for Pain Control,
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 380250
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Group 1 will receive IV acetaminophen 1000mg plus 2 oral capsules "sugar pills" 1 hour prior to surgical incision and 4 hours after initial dose, for a total of two doses of acetaminophen totaling or equaling 2000mg
  Interventions: Drug: IV tylenol 1000mg and 2 oral capsule "sugar pills"
- Group 2 (Experimental): Group 2 will receive an IV "salt water" infusion plus 2 capsules of oral acetaminophen 1 hour prior to surgical incision and 4 hours after initial dose, for a total of two doses totaling or equaling 2000mg.
  Interventions: Drug: 2 capsules Oral Tylenol 2000 mg and IV "salt water"

INTERVENTIONS:
Drug: 2 capsules Oral Tylenol 2000 mg and IV "salt water" — The participants randomized to receive the '2 capsules Oral Acetaminophen 500 mg and IV "salt water repeated 4 hours after that dose to equal 2000mg. A pre-op pain score was obtained and pain scores every 15 min x 1 hour then per recovery routine and they did a 24 hour home diary to record pain scores for 24 hours post surgery. Their opioid morphine equivalent was recorded intraoperatively, recovery and at home. This was compared to the other group receiving IV acetaminophen.and the pain scores and morphine equivalents were collected the same as in the comparative group. Each group received a placebo version oral or iv accordingly.
  Other Names: Acetaminophen is comercially referred to as Tylenol.
  Arms: Group 2
Drug: IV tylenol 1000mg and 2 oral capsule "sugar pills" — IV acetaminophen 1000mg and 2 oral capsule "sugar pills were given to participants that were randomized to receive the IV acetaminophen. The same collection of pain scores and morphine equivalents was completed the same as the other group.
  Other Names: Acetaminophen is comercially referred to as Tylenol.
  Arms: Group 1

SUMMARY:
The purpose of the study is to learn whether perioperative IV (intravenous) administration of acetaminophen (commonly referred to as Tylenol) shows any different clinical outcomes over the oral (by mouth) administration of acetaminophen for a patient having a laparoscopic cholecystectomy. If improved pain scores occur with the administration of IV acetaminophen, it may result in fewer requests for pain-related intervention such as other oral pain medications.

DETAILED DESCRIPTION:
Subjects were enrolled following the listed inclusion and exclusion criteria.

Subjects Eligibility Criteria:

Inclusion Criteria:

Male and female patients ASA I - III . 18 years of age and older

Exclusion Criteria:

Chronic pain syndromes (pain symptoms lasting greater than 3 months), previous abdominal surgery Chronic home narcotic use (patient-reported narcotic use for greater than 3 months) Previous Bowel resection, colon surgery, stomach surgery

. Liver disease (AST or ALT greater than 3 times upper limit of normal), on labs closest to surgical date or within 6 months prior to surgery

Severe renal disease (creatinine clearance less than 30 mL/min), on labs closest to surgical date or within 6 months prior to surgery

Open or emergency surgery (non-scheduled surgery, surgery that must be performed within 6 hours for this particular surgery)

Prior NSAIDS (Non-Steroid Anti-inflammatory Drugs) including COX-2 agents use within the last 24 hours

Use of intraoperative NSAIDs

Contraindication to study drug (including allergic reaction or hypersensitivity to acetaminophen or any of its components;

Taking a medication with known interactions with acetaminophen

Taking chronic oral acetaminophen, greater than 6 months on a daily basis at a dose greater than 3000mg/day

Pregnancy

Current or past alcohol abuse (within the past 2 years)

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ASA I - III (A system used by anesthesiologists to stratify severity of patients' underlying disease and potential for suffering complications from general anesthesia ), 18 years of age and older
* Patient must be scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* Chronic pain syndromes (pain symptoms lasting greater than 3 months), previous abdominal surgery
* Chronic home narcotic use (patient-reported narcotic use for greater than 3 months)
* Liver disease (AST or ALT greater than 3 times upper limit of normal), on labs closest to surgical date or within 6 months prior to surgery
* Severe renal disease (creatinine clearance less than 30 mL/min), on labs closest to surgical date or within 6 months prior to surgery
* Open or emergency surgery (non-scheduled surgery, surgery that must be performed within 6 hours for this particular surgery)
* Prior NSAIDS(Non-Steroid Anti-inflammatory Drugs) including COX-2 agents use within the last 24 hours
* Use of intraoperative NSAIDs
* Contraindication to study drug (including allergic reaction or hypersensitivity to acetaminophen or any of its components;
* On a medication with known interactions with acetaminophen
* On chronic oral acetaminophen, greater than 6 months on a daily basis at a dose greater than 3000mg/day
* Pregnancy
* Current or past alcohol abuse (within the past 2 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Plunkett, MD, Principal Investigator — Womack Army Medical Center
Locations (1):
- Womack Army Medical Center, Fort Bragg, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients (male and non-pregnant females, 18 years of age or older) with symptomatic cholelithiasis and ASA rating of I-III scheduled to undergo elective LapChole were eligible for this trial.
Groups:
- IV Acetaminophen 1000mg + 2 Oral "Sugar Pills": Group 1 will receive IV acetaminophen 1000mg plus 2 oral capsules "sugar pills" 1 hour prior to surgical incision and 4 hours after initial dose, for a total of two doses of acetaminophen totaling or equaling 2000mg
  IV tylenol 1000mg and 2 oral capsule "sugar pills": IV acetaminophen 1000mg and 2 oral capsule "sugar pills were given to participants that were randomized to receive the IV acetaminophen. The same collection of pain scores and morphine equivalents was completed the same as the other group.
- Oral Acetaminophen 2 Capsules + "IV Salt Water": Group 2 will receive an IV "salt water" infusion plus 2 capsules of oral acetaminophen 1 hour prior to surgical incision and 4 hours after initial dose, for a total of two doses totaling or equaling 2000mg.
  2 capsules Oral Tylenol 2000 mg and IV "salt water": The participants randomized to receive the '2 capsules Oral Acetaminophenl 500 mg and IV "salt water repeated 4 hours after that dose to equal 2000mg. A pre-op pain score was obtained and pain scores every 15 min x 1 hour then per recovery routine and they did a 24 hour home diary to record pain scores for 24 hours post surgery. Their opioid morphine equivalent was recorded intraoperatively, recovery and at home. This was compared to the other group receiving IV acetaminophen.and the pain scores and morphine equivalents were collected the same as in the comparative group. Each group received a placebo version oral or iv accordingly.
Period: Overall Study
Arm/Group | IV Acetaminophen 1000mg + 2 Oral "Sugar Pills" | Oral Acetaminophen 2 Capsules + "IV Salt Water"
Started | 34 | 33
Completed | 28 | 22
Not Completed | 6 | 11
Not completed — Lost to Follow-up | 5 | 6
Not completed — didn't qualify | 1 | 2
Not completed — pharmacy error | 0 | 1
Not completed — missed med dose | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 2: Group 2 will receive an IV "salt water" infusion plus 2 capsules of oral acetaminophen 1 hour prior to surgical incision and 4 hours after initial dose, for a total of two doses totaling or equaling 2000mg.
  2 capsules Oral Tylenol 2000 mg and IV "salt water": The participants randomized to receive the '2 capsules Oral Acetaminophenl 500 mg and IV "salt water repeated 4 hours after that dose to equal 2000mg. A pre-op pain score was obtained and pain scores every 15 min x 1 hour then per recovery routine and they did a 24 hour home diary to record pain scores for 24 hours post surgery. Their opioid morphine equivalent was recorded intraoperatively, recovery and at home. This was compared to the other group receiving IV acetaminophen.and the pain scores and morphine equivalents were collected the same as in the comparative group. Each group received a placebo version oral or iv accordingly.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 28 | 22 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 22 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.64 (12.13) | 37.00 (10.65) | 40.32 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 7 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 21 | 16 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 28 | 22 | 50

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: Pain after treatment with IV versus oral tylenol will be assessed via pain scores utilizing an numerical rating scale (NRS) )0-10 with 0 as no pain and 10 as worst pain with 5 as moderate pain and faces accompanied the scores with full smile on no pain to tears and frown on worst pain.
Time Frame: 24 hours after discharge
Measure: Mean (Standard Deviation); unit: NRS scale
Groups:
- Group 1: A Repeated Analyses of Variance was conducted to determine if there were significant differences between the IV and PO groups relative to pain over seven times.
- Group 2: A Repeated Analyses of Variance was conducted to determine if there were significant differences between the IV and PO groups relative to pain over seven times. There were no significant differences between the groups over time, Wilks' Lambda (P = 0.875). (Table 4 and Figure 1)
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 28 | 22
NRS scale
  pre-op | 1.41 (2.09) | 1.73 (1.93)
  Arrival in PACU | 1.61 (2.78) | 2.32 (2.73)
  Discharge from PACU | 2.36 (1.73) | 2.64 (1.56)
  Discharge+6hrs | 4.81 (2.24) | 4.81 (1.69)
  Discharge+12hrs | 5.09 (2.60) | 4.71 (2.08)
  Discharge+18hrs | 4.12 (2.62) | 4.21 (2.07)
  Discharge+24hrs | 3.96 (2.47) | 4.09 (1.77)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority or Other; p = 0.875, Repeated analysis of variance

2. Secondary Outcome: Total Opioid Consumption From Time of First Waking to T24
Description: Pain diary will be filled out every 6 hours for 24 hours after discharge in which the following will be recorded:
  * Opioid consumption from first waking to T4
  * Total opioid consumption from T0 to T4
  * Total opioid consumption from time of first waking to T24
Time Frame: every 6 hours for 24 hours
Measure: Mean (Standard Deviation); unit: milligrams
Groups:
- Group 1: This group consisted of 28 subjects' data that was analyzed. Of the 28 there were 7 males 21 females.
- Group 2: This group consisted of 22 subjects that received the oral acetaminophen and IV placebo. Of the 22 there was 1 male and 21 female.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 28 | 22
milligrams
  PACU | 13.46 (23.20) | 17.41 (17.91)
  Home Consumption | 36.96 (33.19) | 39.56 (37.56)
  Total consumption from peration to 24 hrs | 153.38 (57.32) | 163.86 (78.04)
Statistical Analysis 1: Comparison: Group 1; Test type: Superiority or Other; p > 0.05, Manova

ADVERSE EVENTS:
Time Frame: The adverse event data was collected over the course of the subjects hospital stay starting with the time the subject received his first dose of acetaminophen.
Groups:
- Group 1: .Found to have gangreouns gallbladder and stayed greater 24 hours; upon investigation found not related to the acetaminophen
- Group 2: No adverse events
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/22
Other Adverse Events (participants affected / at risk) | 2/28 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=28) | Group 2 (N=22)
Hospitalization greater 24 hours (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=28) | Group 2 (N=22)
hospitalizatoin (Cardiac disorders) | 1 (1) | 0 (0) — This subject had a planned admit and was in greater than 24 hours after the surgery, she had a cardiac history and was kept as a precaution
ER visit (Renal and urinary disorders) | 1 (1) | 0 (0) — subject came to the ER POD 1 for urinary retention post catheter removal, IRB informed but determined non related. She was sent home again.

LIMITATIONS AND CAVEATS:
Small sample size Only one institution utilized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No